CLINICAL TRIAL: NCT00197483
Title: Effective Adjunctive Use of Pergolide With Risperidone for Cognitive Impairment and Negative Symptoms in Schizophrenia
Brief Title: Effective Adjunctive Use of Pergolide for Cognitive Impairment and Negative Symptoms in Schizophrenia
Status: Suspended | Type: Observational
Sponsor: Hamamatsu University (Other)
Other Study IDs: 01T-080
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Schizophrenia; Negative Symptoms; Cognitive Impairments
Keywords: Pergolide; Dopamine D1; Schizophrenia; Cognitive disturbance; Negative symptoms
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction; Cognition Disorders | interventions — Pergolide; Pharmaceutical Preparations

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Drug: Pergolide (drug)

SUMMARY:
Dopamine has been closely associated with prefrontal function. The hypothesis that a lower dopaminergic activity is associated with negative symptoms and cognitive dysfunction observed in the patients of schizophrenia is of a heuristic value in guiding research in this area. This hypothesis led us to test whether pergolide, a D1/D2 agonist, could improve negative symptoms and cognitive impairments prevailing in most patients with schizophrenia. This double-blind placebo controlled study will investigate the remedial effect of pergolide on negative symptoms and cognitive impairments in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Were age 18-50 years, met the DSM-IV criteria for schizophrenia
* Were treated with a stable dose of risperidone, raging 2 to 6mg, for more than 8 weeks
* Had a score ≥15 on negative subscale items in Positive and Negative Syndrome Scale (PANSS)
* Had a minimum period of symptom stability, defined as no more than 20% change on consecutive ratings on PANSS for at lease 4 weeks

Exclusion Criteria:

* Had a history of medical condition or drug treatment that may have affected cognitive performance
* Had a history of other psychiatric disorders

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 2003-03

CONTACTS AND LOCATIONS:
Overall Officials: Norio Mori, Ph.D, Study Chair — Hamamatsu University, School of Medicine, Department of Psychiatry and Neurology
Locations (1):
- Hamamatsu University Hospital, Hamamatsu, Shizuoka, Japan

REFERENCES:
- [Background] Kimberg DY, D'Esposito M. Cognitive effects of the dopamine receptor agonist pergolide. Neuropsychologia. 2003;41(8):1020-7. doi: 10.1016/s0028-3932(02)00317-2. PMID 12667537
- [Background] Muller U, von Cramon DY, Pollmann S. D1- versus D2-receptor modulation of visuospatial working memory in humans. J Neurosci. 1998 Apr 1;18(7):2720-8. doi: 10.1523/JNEUROSCI.18-07-02720.1998. PMID 9502829
- [Background] Wang M, Vijayraghavan S, Goldman-Rakic PS. Selective D2 receptor actions on the functional circuitry of working memory. Science. 2004 Feb 6;303(5659):853-6. doi: 10.1126/science.1091162. PMID 14764884
- [Background] Goldman-Rakic PS, Castner SA, Svensson TH, Siever LJ, Williams GV. Targeting the dopamine D1 receptor in schizophrenia: insights for cognitive dysfunction. Psychopharmacology (Berl). 2004 Jun;174(1):3-16. doi: 10.1007/s00213-004-1793-y. Epub 2004 Apr 30. PMID 15118803